CLINICAL TRIAL: NCT01000337
Title: The Impact of Sevoflurane and Propofol Anesthesia on Hepatic Apoptosis Markers
Brief Title: Markers of Liver Apoptosis After Anesthesia With Sevoflurane or Propofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Argyro Fassoulaki, MD, PhD, DEAA, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Σ-74/07-07-2009
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2012-09-11 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Liver Dysfunction
Keywords: Liver Apoptosis
MeSH Terms: conditions — Liver Diseases | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sevoflurane (Active Comparator): Volatile anesthetic
  Interventions: Drug: Sevoflurane
- Propofol (Active Comparator): Intravenous anesthetic
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane concentration for induction of anesthesia 7-8%, for maintenance of anesthesia 2%.
  Other Names: Sevorane, 2802252901023,
  Arms: sevoflurane
Drug: Propofol — Propofol to induce anesthesia 2.5 mg/kg, for maintenance of anesthesia 6 mg/kg/h
  Other Names: Lipuro, 2802467102017
  Arms: Propofol

SUMMARY:
Anesthesia may affect the function of vital organs. Liver is one of them. The investigator's hypothesis is that intravenous or inhalation anesthesia does not impair liver function as assessed by more elegant tests like markers indicating liver apoptosis. In the present randomized prospective trial female patients scheduled for mastectomy or thyroidectomy will receive inhalation or total intravenous anesthesia and markers for liver dysfunction will be determined.

DETAILED DESCRIPTION:
Female patients undergoing mastectomy or thyroidectomy under sevoflurane or propofol anesthesia will be recruited for the study. The type of anesthesia will be determined in a random way using a computer generated table.

All patients will be preoxygenated for 3 minutes before induction of anesthesia. Patients assigned to the sevoflurane group will receive an inhalation induction with sevoflurane via a primed anesthetic circle system and anesthesia will be maintained with sevoflurane. In the propofol group patients anaesthesia will be induced and maintained with propofol.

Blood samples for liver apoptotic markers will be collected before induction of anesthesia, after skin closure as well as 24 and 48 hours postoperatively.

Blood samples will be centrifuged, stored at -80 degrees Celsius and analyzed for M30 and M60 values with radioimmunoassay technique. Serum glutamic pyruvic transaminase (SGPT) and serum glutamic oxaloacetic transaminase (SGOT) levels will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 30 and 65 years old scheduled for thyroidectomy or breast surgery for cancer

Exclusion Criteria:

* Drug intake which may affect liver function
* Severe cardiovascular or respiratory disease
* Hepatic or renal dysfunction
* Pregnancy
* Alcohol and drug abuse
* Body Mass Index (BMI) > 35

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Argyro Fassoulaki, MD,PhD,DEAA, Study Chair — Chairman Department of Anesthesiology, Aretaieio Hospital
Locations (1):
- Aretaieio Hospital, University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between October 2009 and July 2011 in Aretaieo University Hospital, Athens, Greece
Pre-assignment Details: Potential participants prior to group assignment were enrolled but excluded from the trial due to exclusion criteria as defined by the study protocol
Groups:
- Sevoflurane: Volatile anesthetic used to induce and maintain general anaeshesia. To induce anaesthesia the inspired concentration recommended is 8% in oxyfen to maintain anaesthesia the inspired concentration is 1-2%. The drug is administered continuously during surgery using a specially designed vaporizer. The depth of anesthesia obtained during sevoflurane administration is monitored by the end expired concentration of sevoflurane and by the bispectral index monitoring. The effect of sevoflurane on the liver for the predetermined clinically applicable concentrations was evaluated.
- Propofol: Intravenous anesthetic suitable for induction and maintainance of general anesthesia. Anaesthesia is induced by administereing intravenously 2-2.5 mg/kg body weight and maintained by continuous intravenous infusion of 6 mg/kg/hour of propofol by means of an electric infusion pump.
  The depth of anesthesia during propofol anesthesia is monitored by the bispectral index monitoring. The effect of propofol on the liver for the predetermined clinically applicable concentrations was evaluated.
Period: Overall Study
Arm/Group | Sevoflurane | Propofol
Started | 34 | 33
Completed | 30 | 30
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevoflurane | Propofol | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 33 | 67
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.93 (10.19) | 48.30 (10.81) | 51.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Greece | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Changes in the M30 and M65 Markers Related to the Anesthesia Type
Description: Blood samples for determination of the markers M30 and M65 as well as the serum transaminases were collected preoperatively, at the end of surgery, 24 and 48 hours postoperatively.
Time Frame: preoperatively, end of surgery, 24 and 48 hours postoperatively
Population: For an effect size of 0.20 assuming a two-sided error type I error of 0.05 and a power of 0.80, a sample size of 60 sixty patients (30 patients in each group) would be required.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Sevoflurane | Propofol
Number analyzed (Participants) | 34 | 33
U/L
  M30 marker preoperatively | 237.27 (95.46) | 279.97 (228.96)
  M65 marker preoperatively | 427.33 (225.70) | 470.30 (261.98)
  M30 marker postoperatively | 241.83 (108.60) | 299.97 (243.85)
  M65 marker postoperatively | 480.90 (227.51) | 478.27 (271.53)
  M30 marker 24h postoperatively | 231.10 (93.67) | 267.17 (197.66)
  M65 marker 24h postoperatively | 389.17 (158.12) | 456.43 (338.91)
  M30 marker 48h postoperatively | 234.10 (127.27) | 254.20 (188.61)
  M65 marker 48h postoperatively | 404.20 (144.01) | 485.53 (272.56)

2. Secondary Outcome: Transaminases
Time Frame: February 2011
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the first 48 hours after surgery
Arm/Group | Sevoflurane | Propofol
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33

LIMITATIONS AND CAVEATS:
The study was accomplished with no problems leading to data questioning.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No